CLINICAL TRIAL: NCT07121738
Title: A Prospective Study of a Lifestyle Medicine Survivorship Program for Patients With Gynecologic Cancer
Acronym: HEAL-GYN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Collaborators: State of Florida Department of Health (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2337720
Record Dates: First submitted 2025-08-07; First posted 2025-08-13 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Gynecologic Cancers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral (Experimental): Evidence-based lifestyle medicine program for cancer survivors
  Interventions: Behavioral: Healthy Eating Active Lifestyle (HEAL): Gyn Cancer Program

INTERVENTIONS:
Behavioral: Healthy Eating Active Lifestyle (HEAL): Gyn Cancer Program — Evidence-based lifestyle medicine program for cancer survivors

SUMMARY:
This study will examine the effects of an 8-week intervention called the Healthy Eating Active Lifestyle (HEAL)-GYN program on participants' 1) self-efficacy 2) lifestyle factors, including physical activity and diet, as well as mental health and overall well-being, and 3) biometrics and biomarkers.

DETAILED DESCRIPTION:
This study will examine the effects of an 8-week intervention called the Healthy Eating Active Lifestyle (HEAL)-GYN program. This telemedicine-based rehabilitation course for patients with gynecologic cancer focuses on lifestyle changes in exercise, nutrition, sleep, social integration, stress management, and avoidance of risk behaviors, such as smoking and alcohol. Led by a certified lifestyle medicine oncologist, the multidisciplinary program includes personalized goal-setting and experiential instruction on these topics. A prospective study will be conducted with up to 64 participants who are patients with gynecologic cancer to examine the effects of the HEAL-GYN program on 1) self-efficacy 2) lifestyle factors, including physical activity and diet, as well as mental health and overall well-being, and 3) biometrics and biomarkers. Participants will complete a survey package at baseline, endpoint, 1-month follow-up, and 3-month follow-up timepoints, which includes the following validated instruments: Weight Efficacy Lifestyle Questionnaire, Godin-Shephard Leisure-Time Physical Activity Questionnaire, Diet History Questionnaire III, Pittsburgh Sleep Quality Index, Body Image Scale, Perceived Stress Scale, Generalized Anxiety Disorder 7-item scale (GAD-7), Patient Health Questionnaire 9-item scale (PHQ-9), and Functional Assessment of Cancer Therapy - General. Objective measurements of physical activity and sleep will be collected using a wearable activity tracker. During home health visits, data related to biometrics will be collected, along with basic lab values and biomarkers of adiponectin, insulin sensitivity, and inflammatory markers through blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years old or over
* Diagnosis of gynecologic cancer
* Current patient in the Central Florida area
* Completing or have completed chemotherapy treatment within approximately the past 3 months before starting the program
* Able to speak, read, and understand the English language.

Exclusion Criteria:

* Not willing or able to provide informed consent
* Not willing or able to comply with all study procedures and requirement for the duration of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Weight Efficacy Lifestyle (WEL) Questionnaire | Baseline, Endpoint (week 8), 1-month follow-up, 3-month follow up
  A 20-item questionnaire measuring eating self-efficacy across five domains: negative emotions, availability, social pressure, physical discomfort, and positive activities. Each item is rated on a 10-point scale (0 = Not confident, 9 = Very confident) for the participant's ability to resist overeating in various situations. Higher scores indicate greater confidence in managing eating behaviors (higher eating self-efficacy).

SECONDARY OUTCOMES:
Godin-Shephard Leisure-Time Physical Activity Questionnaire | Baseline, Endpoint (week 8), 1-month follow-up, 3-month follow up
  A 3-item self-report questionnaire asking the number of times per week one engages in strenuous, moderate, and mild leisure exercise. Participants enter frequency counts for each category, which are used to compute a weekly activity score. Higher scores indicate higher physical activity level.
Diet History Questionnaire III (DHQ III) | Baseline, Endpoint (week 8), 1-month follow-up, 3-month follow up
  A ~130-item food frequency questionnaire collecting dietary intake information. Participants report how often they consume various foods and beverages and sometimes portion size. It measures habitual dietary intake and nutrient consumption patterns.
Pittsburgh Sleep Quality Index (PSQI) | Baseline, Endpoint (week 8), 1-month follow-up, 3-month follow up
  A 19-item questionnaire assessing habitual sleep quality over the past month in terms of bedtime, sleep latency, duration, efficiency, disturbances, use of sleep aids, and daytime dysfunction. Each item is rated on a 4-point scale (0 = Not during the past month to 3 = ≥3 times/week). A total score is computed (0-21). Higher scores indicate poorer sleep quality.
Body Image Scale | Baseline, Endpoint (week 8), 1-month follow-up, 3-month follow up
  A 10-item self-report scale developed for cancer patients to evaluate body image changes. Each item is rated on a 4-point scale (0 = Not at all to 3 = Very much). A total score is computed (0-30). Higher scores indicate greater body image disturbance or dissatisfaction.
Perceived Stress Scale | Baseline, Endpoint (week 8), 1-month follow-up, 3-month follow up
  A 10-item scale assessing the degree to which situations in one's life are appraised as stressful. Each item is rated from on a 5-point scale (0 = Never to 4 = Very Often) based on the frequency of feelings in the past month. A total score is computed (0-40). Higher scores indicate higher stress.
Generalized Anxiety Disorder - 7-item scale (GAD-7) | Baseline, Endpoint (week 8), 1-month follow-up, 3-month follow up
  A 7-item screening questionnaire for generalized anxiety. Each item is rated on a 4-point scale (0 = Not at all to 3 = Nearly every day) for how often it occurred over the last 2 weeks. A total score is computed (0-21). Higher totals indicate more severe anxiety symptoms.
Patient Health Questionnaire - 9-item scale (PHQ-9) | Baseline, Endpoint (week 8), 1-month follow-up, 3-month follow up
  A 9-item depression screening tool. Each item is rated on a 4-point scale (0 = Not at all to 3 = Nearly every day) for how often it occurred over the last 2 weeks. A total score is computed (0-27). Higher totals indicate more severe depressive symptoms.
Functional Assessment of Cancer Therapy - General (FACT-G) | Baseline, Endpoint (week 8), 1-month follow-up, 3-month follow up
  A 27-item validated questionnaire measuring health-related quality of life in cancer patients across four domains: physical, social/family, emotional, and functional. Each item is rated on a 5-point scale (0 = Not at all to 4 = Very much). Domain scores are summed to calculate a total score. Higher scores indicate better quality of life.
Height | Baseline, 3-month follow up
  Participant's standing height, measured in inches using a stadiometer or measuring tape.
Weight | Baseline, 3-month follow up
  Participant's body weight, measured in pounds using a scale
Waist-to-hip ratio | Baseline, 3-month follow up
  Ratio of waist circumference to hip circumference, both measured in inches using a tape measure.
Basic lab values | Baseline, 3-month follow up
  Comprehensive Metabolic Panel; Blood lipid panel including Low-Density Lipoprotein (LDL), High-Density Lipoprotein (HDL), and triglycerides; Hemoglobin A1c;
Adiponectin | Baseline, 3-month follow up
  A blood biomarker (hormone), measured via blood sample.
Insulin sensitivity | Baseline, 3-month follow up
  An index of how responsive the body is to insulin, measured via blood sample.
Inflammatory markers | Baseline, 3-month follow up
  Includes C-reactive protein (CRP), Interleukin-6 (IL-6), and Tumor Necrosis Factor-alpha (TNF-α), measured via blood sample.
Physical activity minutes | Baseline, Endpoint (week 8), 1-month follow-up, 3-month follow up
  Objective measurement of daily minutes spent in light, moderate, and vigorous activity using a wearable activity tracker.
Sleep minutes | Baseline, Endpoint (week 8), 1-month follow-up, 3-month follow up
  Objective measurement of nightly minutes spent in light, deep, and REM sleep stages using a wearable activity tracker.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda T Sawyer, PhD, Principal Investigator — AdventHealth
Locations (1):
- AdventHealth, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McKenzie ND, Ahmad S. Impact of Lifestyle Interventions on Gynecologic Cancers: Beyond Diet and Exercise. Am J Lifestyle Med. 2022 Sep 14;18(1):7-20. doi: 10.1177/15598276221123764. eCollection 2024 Jan-Feb. PMID 39184272
- [Background] Clark MM, Abrams DB, Niaura RS, Eaton CA, Rossi JS. Self-efficacy in weight management. J Consult Clin Psychol. 1991 Oct;59(5):739-44. doi: 10.1037//0022-006x.59.5.739. PMID 1955608
- [Background] Godin G. The Godin-Shephard Leisure-Time Physical Activity Questionnaire. Health Fitness J Can. 2011;4(1):18-22. doi:10.14288/hfjc.v4i1.82
- [Background] Thompson FE, Subar AF, Brown CC, Smith AF, Sharbaugh CO, Jobe JB, Mittl B, Gibson JT, Ziegler RG. Cognitive research enhances accuracy of food frequency questionnaire reports: results of an experimental validation study. J Am Diet Assoc. 2002 Feb;102(2):212-25. doi: 10.1016/s0002-8223(02)90050-7. PMID 11846115
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Hopwood P. The assessment of body image in cancer patients. Eur J Cancer. 1993;29A(2):276-81. doi: 10.1016/0959-8049(93)90193-j. PMID 8422297
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Webster K, Cella D, Yost K. The Functional Assessment of Chronic Illness Therapy (FACIT) Measurement System: properties, applications, and interpretation. Health Qual Life Outcomes. 2003 Dec 16;1:79. doi: 10.1186/1477-7525-1-79. PMID 14678568
- [Background] Victorson D, Barocas J, Song J, Cella D. Reliability across studies from the functional assessment of cancer therapy-general (FACT-G) and its subscales: a reliability generalization. Qual Life Res. 2008 Nov;17(9):1137-46. doi: 10.1007/s11136-008-9398-2. Epub 2008 Oct 8. PMID 18841493